CLINICAL TRIAL: NCT03611894
Title: Comparison of the Radiological Pattern Between the Cerebral Stroke of Arterial and Venous Origin
Acronym: PATTERN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2017_843_0035
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Stroke; Superior Sagittal Sinus Thrombosis; Venous Thromboses
Keywords: RMI
MeSH Terms: conditions — Stroke; Sagittal Sinus Thrombosis; Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- hemorrhagic ischemia: comparison between clinical characteristics and the confirmed diagnosis by RMI (magnetic resonance Imaging)
  Interventions: Other: radiological comparison
- nonhemorrhagic ischemia: comparison between clinical characteristics and the confirmed diagnosis by RMI (magnetic resonance Imaging)
  Interventions: Other: radiological comparison
- intracerebral hematoma: comparison between clinical characteristics and the confirmed diagnosis by RMI (magnetic resonance Imaging)
  Interventions: Other: radiological comparison

INTERVENTIONS:
Other: radiological comparison — comparison between clinical and radiological characteristics

SUMMARY:
There are few published data on the patterns of parenchymal imaging abnormalities in a context of cerebral venous thrombosis (CVT). The objectives of the present study were to describe the patterns of parenchymal lesions associated with CVT and to determine the lesion sites.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patients with CVT
* parenchymal lesions on magnetic resonance imaging

Exclusion Criteria:

* No CVT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators want to include consecutively hospitalized patients with CVT and parenchymal lesions on magnetic resonance imaging.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
patterns | 0
  describe the patterns of parenchymal lesions associated with CVT and to determine the lesion sites.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Arnoux, MD, Principal Investigator — CHU Amiens
Locations (2):
- France (2):
  - CHU Amiens, Amiens
  - CHU Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No